CLINICAL TRIAL: NCT01808612
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind, Parallel-Design Study to Evaluate the Short-Term, Fixed Dose Efficacy and Safety of LY110140 Once Daily Dosing in Japanese Patients With Major Depressive Disorder
Brief Title: A Study of Fluoxetine in Major Depressive Disorder (MDD) Short-Term Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14595; B1Y-JE-HCLV (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg Fluoxetine (Experimental): 20 milligrams (mg) fluoxetine (capsules) administered orally, once daily, for 6 weeks
  Interventions: Drug: Fluoxetine
- 40 mg Fluoxetine (Experimental): 40 mg fluoxetine (capsules) administered orally, once daily, for 6 weeks
  Interventions: Drug: Fluoxetine
- Placebo (Placebo Comparator): Placebo (capsules) administered orally, once daily, for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine
  Other Names: LY110140; Fluoxetine Hydrochloride; Prozac; Sarafem
  Arms: 20 mg Fluoxetine; 40 mg Fluoxetine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the short-term efficacy and safety of Fluoxetine in Japanese adult participants with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient Japanese participants diagnosed with MDD
* Diagnosis of moderate or greater severity of MDD
* Agree to abstain from sexual activity or to use a reliable method of birth control
* Judged to be reliable (agree to keep appointments for clinic visits and to undergo all tests and examinations required by the protocol)

Exclusion Criteria:

* Have previously been exposed to fluoxetine (LY110140) for any indication in the past
* Significant suicidal risk
* Have a current or previous diagnosis of bipolar disorder, psychotic depression, schizophrenia or other psychotic disorder, anorexia, bulimia, obsessive compulsive disorder, or post-traumatic stress disorder
* Have a history of substance abuse or dependence within the past 6 months, excluding caffeine and nicotine
* Have initiated, stopped, or changed the type or intensity of psychotherapy within 6 weeks
* Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), or vagus nerve stimulation (VNS) within 1 year
* Have had treatment with a Monoamine oxidase inhibitor (MAOI) within 14 days
* Need to use thioridazine or pimozide during the study
* Have previously enrolled, completed, or withdrawn from this study
* Have a positive urine drug screen for drugs with abuse potential
* Female participants who are either pregnant, nursing, or have recently given birth, or male participants who are planning for their partners to be or become pregnant
* Have a history of seizure disorder
* Have frequent or severe allergic reactions to multiple medications
* Have a serious or unstable medical illness or condition, or psychological condition
* Participants deemed ineligible by the investigator or sub-investigator for other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- Japan (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shiga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 3 periods: a single-blind screening period (1 week of placebo), a double-blind short-term treatment period (1 week of placebo followed by randomization in a 2:1:3 fashion to 20 milligrams [mg] fluoxetine, 40 mg fluoxetine, or placebo, respectively, for 6 weeks), and a single-blind discontinuation period (2 weeks of placebo).
Groups:
- 20 mg Fluoxetine: Treatment Period: 20 milligrams (mg) fluoxetine (capsules) administered orally, once daily, for 6 weeks
  Discontinuation Period: placebo (capsules) administered orally, once daily, for 2 weeks
- 40 mg Fluoxetine: Treatment Period: 40 mg fluoxetine (capsules) administered orally, once daily, for 6 weeks
  Discontinuation Period: placebo (capsules) administered orally, once daily, for 2 weeks
- Placebo: Treatment Period: placebo (capsules) administered orally, once daily, for 6 weeks
  Discontinuation Period: placebo (capsules) administered orally, once daily, for 2 weeks
Period: Treatment Period
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Started | 169 | 84 | 260
Received at Least 1 Dose of Study Drug | 168 (Only these participants were included in the study analyses (ie, Full Analysis Set).) | 83 (Only these participants were included in the study analyses (ie, Full Analysis Set).) | 259 (Only these participants were included in the study analyses (ie, Full Analysis Set).)
Completed | 154 (67 participants who completed the Treatment Period did not enter the Discontinuation Period.) | 77 (39 participants who completed the Treatment Period did not enter the Discontinuation Period.) | 246 (101 participants who completed the Treatment Period did not enter the Discontinuation Period.)
Not Completed | 15 | 7 | 14
Not completed — Adverse Event | 8 | 4 | 3
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 4
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 2
Period: Discontinuation Period
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Started | 87 | 38 | 145
Completed | 85 | 37 | 145
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- 20 mg Fluoxetine: 20 mg fluoxetine (capsules) administered orally, once daily, for 6 weeks
- Total: Total of all reporting groups
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo | Total
Number analyzed (Participants) | 168 | 83 | 259 | 510
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.05 (11.19) | 39.58 (10.56) | 38.54 (11.65) | 39.20 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 33 | 129 | 245
  Male | 85 | 50 | 130 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 168 | 83 | 259 | 510
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 168 | 83 | 259 | 510
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 168 | 83 | 259 | 510

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to 6-Week Endpoint on the 21-Item Hamilton Depression Rating Scale (HAMD21) Total Score
Description: HAMD21 is a 21-item assessment used to measure depression severity. Items were rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score ranging from 0 (not at all depressed) to 64 (severely depressed). Least squares (LS) means were calculated using mixed-model repeated measures (MMRM) adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline HAMD21 total score.
Time Frame: Baseline, 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 total score during the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 259
units on a scale | -6.18 (0.57) | -6.25 (0.77) | -6.91 (0.49)
Statistical Analysis 1: Comparison: 20 mg Fluoxetine vs Placebo; Approximately 522 participants were to be enrolled. Randomization was to be 2:1:3 (20 mg fluoxetine:40 mg fluoxetine:placebo). Assuming 5% of participants would have missing post-baseline data, the study had 85% power to detect an effect size of 0.33 (20 mg fluoxetine compared to placebo on HAMD21 total score) based on simulations with a 0.05 two-sided significance level; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis; LS Mean Difference = 0.73, 95% CI 2-sided [-0.55 to 2.00]

2. Secondary Outcome: Mean Change From Baseline to 6-Week Endpoint on the HAMD21 Subscale Scores
Description: HAMD17 total scores and subscale scores from the HAMD21 are presented. HAMD17 is a 17-item assessment of depression severity (total scores range from 0-52). The Maier subscale (Items 1, 2, 7-10) represents the core symptoms of depression (0-24). Anxiety/Somatization subscale (Items 10-13, 15, 17) evaluates severity of psychic and somatic manifestations of anxiety as well as agitation (0-18). Retardation/Somatization subscale (Items 1, 7, 8, 14) evaluates dysfunction in mood, work, and sexual activity, as well as overall motor retardation (0-14). Sleep subscale (Items 4-6) assesses insomnia (0-6). Individual item scores may range from 0-4 or 0-2. Higher scores indicate more severe symptoms. LS means were calculated using MMRM adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline score.
Time Frame: Baseline, 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 subscale score during the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 259
units on a scale
  HAMD17 total score | -5.59 (0.53) | -5.61 (0.71) | -6.27 (0.45)
  Maier subscale score | -3.35 (0.30) | -3.39 (0.40) | -3.30 (0.26)
  Anxiety/Somatization subscale score | -2.04 (0.21) | -1.84 (0.28) | -2.06 (0.18)
  Retardation/Somatization subscale score | -2.00 (0.20) | -2.21 (0.27) | -2.23 (0.17)
  Sleep subscale score | -0.83 (0.15) | -0.81 (0.20) | -1.10 (0.13)

3. Secondary Outcome: Percentage of Participants Achieving a Response at 6-Week Endpoint
Description: The percentage of participants achieving a response (defined as a ≥50% improvement from baseline on the HAMD21 total score) was calculated by dividing the number of participants achieving a response at last observation by the total number of participants at risk, multiplied by 100.
Time Frame: up to 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline HAMD21 total score during the Treatment Period. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 259
percentage of participants | 23.8 | 18.1 | 27.8

4. Secondary Outcome: Percentage of Participants Achieving a Remission at 6-Week Endpoint
Description: The percentage of participants achieving a remission (defined as a HAMD21 total score ≤7) was calculated by dividing the number of participants achieving a remission at last observation by the total number of participants at risk, multiplied by 100.
Time Frame: up to 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline (which had not achieved remission threshold criteria) and had at least 1 post-baseline HAMD21 total score during the Treatment Period. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 258
percentage of participants | 9.5 | 9.6 | 15.1

5. Secondary Outcome: Mean Change From Baseline to 6-Week Endpoint on the Clinical Global Impression of Severity (CGI-S) Scale
Description: CGI-S measures severity of illness at the time of assessment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). LS means were calculated using MMRM adjusting for the random effect of participant and fixed categorical effects of treatment, pooled investigative site, visit, and treatment-by-visit interaction, as well as the continuous fixed covariate of baseline CGI-S score.
Time Frame: Baseline, 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline CGI-S score during the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 259
units on a scale | -0.69 (0.08) | -0.67 (0.11) | -0.81 (0.07)

6. Secondary Outcome: Mean Change From Baseline to 6-Week Endpoint in Sheehan Disability Scale (SDS) Total Score and Subscale Scores
Description: SDS was completed by the participant and was used to assess the effect of the participant's symptoms on their work/school (Item 1), social life/leisure activities (Item 2), and family life/home responsibilities (Item 3). Each item was measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total score was the sum of the 3 items and ranged from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. LS means were calculated using analysis of covariance (ANCOVA) adjusting for treatment, pooled investigative site, and baseline SDS score.
Time Frame: Baseline, up to 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with a baseline and at least 1 post-baseline SDS score during the Treatment Period. Missing endpoints were imputed with the last observation carried forward (LOCF) method, using only postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 167 | 81 | 259
units on a scale
  Total score (n=167, 81, 259) | -1.76 (0.59) | -1.55 (0.78) | -1.99 (0.53)
  Work/School subscale score (n=143, 64, 226) | -0.79 (0.27) | -0.34 (0.36) | -0.88 (0.24)
  Social/Leisure subscale score (n=167, 81, 259) | -0.66 (0.23) | -0.81 (0.30) | -0.70 (0.21)
  Family/Home subscale score (n=167, 81, 259) | -0.47 (0.21) | -0.30 (0.28) | -0.41 (0.19)

7. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Collected by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline through 6 weeks
Population: Randomized participants who received at least 1 dose of study drug with at least 1 post-baseline C-SSRS score during the Treatment Period.
Measure: Number; unit: participants
Arm/Group | 20 mg Fluoxetine | 40 mg Fluoxetine | Placebo
Number analyzed (Participants) | 168 | 83 | 259
participants
  Suicidal behavior | 0 | 0 | 1
  Suicidal ideation | 5 | 6 | 8

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were reported for all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo (Treatment Period): Adverse events (AEs) which occurred during the Treatment Period for participants who received placebo administered orally, once daily, for 6 weeks during the Treatment Period
- 20 mg Fluoxetine (Treatment Period): AEs which occurred during the Treatment Period for participants who received 20 mg fluoxetine administered orally, once daily, for 6 weeks during the Treatment Period
- 40 mg Fluoxetine (Treatment Period): AEs which occurred during the Treatment Period for participants who received 40 mg fluoxetine administered orally, once daily, for 6 weeks during the Treatment Period
- Placebo (Discontinuation From Placebo): AEs which occurred during the Discontinuation Period for participants who received placebo during the Treatment Period and who received placebo administered orally, once daily, for 2 weeks during the Discontinuation Period
- Placebo (Discontinuation From 20 mg Fluoxetine): AEs which occurred during the Discontinuation Period for participants who received 20 mg fluoxetine during the Treatment Period and who received placebo administered orally, once daily, for 2 weeks during the Discontinuation Period
- Placebo (Discontinuation From 40 mg Fluoxetine): AEs which occurred during the Discontinuation Period for participants who received 40 mg fluoxetine during the Treatment Period and who received placebo administered orally, once daily, for 2 weeks during the Discontinuation Period
Arm/Group | Placebo (Treatment Period) | 20 mg Fluoxetine (Treatment Period) | 40 mg Fluoxetine (Treatment Period) | Placebo (Discontinuation From Placebo) | Placebo (Discontinuation From 20 mg Fluoxetine) | Placebo (Discontinuation From 40 mg Fluoxetine)
Serious Adverse Events (participants affected / at risk) | 2/259 | 0/168 | 0/83 | 1/145 | 0/87 | 0/38
Other Adverse Events (participants affected / at risk) | 75/259 | 49/168 | 30/83 | 5/145 | 5/87 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (Treatment Period) (N=259) | 20 mg Fluoxetine (Treatment Period) (N=168) | 40 mg Fluoxetine (Treatment Period) (N=83) | Placebo (Discontinuation From Placebo) (N=145) | Placebo (Discontinuation From 20 mg Fluoxetine) (N=87) | Placebo (Discontinuation From 40 mg Fluoxetine) (N=38)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infertility male (Reproductive system and breast disorders) | 1/130 (1) | 0/85 (0) | 0/50 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (Treatment Period) (N=259) | 20 mg Fluoxetine (Treatment Period) (N=168) | 40 mg Fluoxetine (Treatment Period) (N=83) | Placebo (Discontinuation From Placebo) (N=145) | Placebo (Discontinuation From 20 mg Fluoxetine) (N=87) | Placebo (Discontinuation From 40 mg Fluoxetine) (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (17) | 6 (7) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram st segment depression (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endoscopy large bowel (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Qrs axis abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anterograde amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impatience (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/129 (1) | 1/83 (2) | 0/33 (0) | 0 (0) | 0 (0) | 0 (0)
Ejaculation delayed (Reproductive system and breast disorders) | 0/130 (0) | 0/85 (0) | 1/50 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days